CLINICAL TRIAL: NCT00580424
Title: The Effect of Oral Norethindrone on Coagulation Parameters in Women at Increased Risk for Venous Thromboembolic Events
Brief Title: The Effect of the Mini-pill on Blood Factors in Women at Increased Risk for Forming Blood Clots
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Kristen Wright, MD, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08-002
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2007-12

CONDITIONS: Women's Health; Blood Coagulation Disorders
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Norethindrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Norethindrone — Norethindrone 0.35 mg orally daily
  Other Names: Minipill

SUMMARY:
We propose a prospective cohort study to assess the effect of the progesterone only contraceptive pill (minipill) on coagulation parameters known to be associated with risk of thrombosis (blood clots) in women who are at increased risk for forming blood clots. We plan to recruit women with a history of venous thromboembolism (VTE, blood clot in a vein) and women with a history of blood tests which demonstrate an increased risk of thrombosis who desire contraception.

Women enrolled in this study will undergo phlebotomy (blood draw) at baseline (prior to starting the minipill), one and three months. Stored samples will be used to measure D-dimer, C-reactive protein (CRP), antithrombin (AT), factor VIII, free and total protein S, fibrinogen, von Willebrand factor (vWF) and normalized activated protein C sensitivity ratio (nAPCsr). Both groups will undergo a general physical and GYN exam prior to enrollment. This exam and the blood testing will be provided free of charge. Patients will not be prescribed the minipill after completion of the study and will be advised to consult with their primary care physician or hematologist if they wish to continue this medication.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of venous thromboembolism (VTE, blood clot in a vein) and women with a history of blood tests which demonstrate an increased risk of thrombosis who desire contraception.
* Blood tests which demonstrate an increased risk of thrombosis include the following:

  * Hyperhomocysteinemia/MTHFR mutation
  * Prothrombin gene mutation
  * Factor V Leiden heterozygotes
  * Factor V Leiden homozygotes, antithrombin III mutation
  * Protein S deficiency and Protein C deficiency.

Exclusion Criteria:

* Women on current anticoagulation therapy
* Women with a history of oral contraceptive related thrombotic events
* Active or history of cigarette smoking within the past 6 months
* Pregnancy
* Active lactation
* Known hypersensitivity to progestin
* Any history of malignancy
* History within the last three months of surgery or planning surgery during the study period
* Undiagnosed vaginal bleeding
* Active liver disease and history within the last 5 years of alcoholism or drug abuse.
* Additionally, women must be greater than 3 months postpartum and have had two months without contraceptive hormones (such as the birth control pill) and 6 months without Depo-Provera use prior to enrollment.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-12; Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study will be change in coagulation parameters. The proposed sample size of 20 subjects was derived based on having sufficient power to detect a 40% change in the variable D-dimer, a lab measurement. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristen P Wright, MD, Principal Investigator — University of Vermont; Julia V Johnson, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States